CLINICAL TRIAL: NCT01829971
Title: A Multicenter Phase I Study of MRX34, MicroRNA miR-RX34 Liposomal Injection
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Five immune related serious adverse events
Sponsor: Mirna Therapeutics, Inc. (Industry)
Collaborators: Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRX34-101
Record Dates: First submitted 2013-04-08; First posted 2013-04-11 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Primary Liver Cancer; SCLC; Lymphoma; Melanoma; Multiple Myeloma; Renal Cell Carcinoma; NSCLC
Keywords: microRNA; Advanced cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Lymphoma; Melanoma; Multiple Myeloma; Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MRX34 (Experimental): Single agent MRX34
  Interventions: Drug: MRX34

INTERVENTIONS:
Drug: MRX34 — micro RNA therapy

SUMMARY:
This is a study to evaluate the safety of MRX34 in patients with primary liver cancer or other selected solid tumors or hematologic malignancies. The drug is given intravenously, for 5 days in a row and then two weeks off.

DETAILED DESCRIPTION:
This is a Phase I, open-label, multicenter, dose-escalation study to investigate the safety, Pharmacokinetics and Pharmacodynamics of the micro ribonucleic acid (microRNA) MRX34, in patients with unresectable primary liver cancer or advanced or metastatic cancer with or without liver involvement or hematologic malignancies. MRX34 will be administered daily x 5 with 2 weeks off (total of 21 days) for 3 cycles followed by a no-treatment observation period.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years
2. Patients with histologically confirmed viral related hepatocellular, SCLC, non-cutaneous/ non-uveal melanoma, ovarian, TNBC, Sarcoma, Bladder and RCC.
3. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
4. Acceptable liver function:

   * Total bilirubin ≤ 1.5 times the upper limit of normal (ULN); for patients with hepatocellular carcinoma only, total bilirubin ≤ 3 mg/dL (i.e. Child-Pugh Score for bilirubin is no greater than 2).
   * Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase (ALP) ≤ 5 x ULN.
5. Acceptable renal function:

   • Serum creatinine ≤ 1.5 times the ULN, or calculated creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above 1.5 times the institutional normal
6. Acceptable hematological status:

   * Absolute Neutrophil Count (ANC) ≥ 1500 cells/mm3
   * Platelet count ≥ 100,000 plts/mm3 (without transfusion); ≥ 75,000 plts/mm3 for patients with hepatocellular carcinoma only. For hematologic malignancy patients blood counts cited above do not apply
   * Hemoglobin ≥ 9 g/dL
   * For the hematologic malignancy patients, blood count values cited above do not apply.
7. Prothrombin time (PT) or International Normalized Ratio (INR) ≤ 1.25 x ULN; for patients with hepatocellular carcinoma only, INR <1.7 or prothrombin time (PT) or < 4 seconds above ULN (i.e. Child-Pugh Score is no greater than 1 for the coagulation parameter); for patients with hepatocellular carcinoma only, serum albumin > 2.8 g/dL (i.e. Child-Pugh Score for albumin is no greater than 2). For the hematologic malignancy patients, the coagulation and albumin status cited above do not apply
8. For patients with hepatocellular carcinoma only, Child-Pugh Class A (score 5-6) disease. Score for hepatic encephalopathy must be 1; the score for ascites must be no greater than 2 and clinically irrelevant; for the determination of the Child-Pugh Class.

Exclusion Criteria:

1. Myocardial infarction within the past 6 months, unstable and/or symptomatic arrhythmia, or evidence of ischemia on ECG.
2. Active, uncontrolled bacterial, viral, or fungal infections requiring systemic therapy.
3. Pregnant or nursing women.
4. Known infection with human immunodeficiency virus (HIV).
5. Serious nonmalignant disease (e.g., hydronephrosis, liver failure, heart failure, or other conditions) that could compromise protocol objectives in the opinion of the investigator and/or the sponsor.
6. Patients with recent history of hemorrhage and patients predisposed to hemorrhage due to coagulopathies or structural anomalies.
7. Patients who require treatment with therapeutic doses of coumadin-type anticoagulants (maximum daily dose of 1mg allowed for port line patency permitted).
8. Patients with cirrhosis classed as Child-Pugh B or C.
9. Patients with central nervous system (CNS) metastasis. Intrathecal chemotherapy is allowed for patients who require CNS prophylaxis or therapy.
10. Patients for whom dexamethasone is contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2013-04; Primary Completion 2017-03 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD) for MRX34 and the recommended phase 2 dose (RPh2D) | 18 months
  Dose-limiting toxicity (DLT) in 3-6 patients at the end of one treatment cycle

SECONDARY OUTCOMES:
Peak blood concentration and Area Under the Curve (AUC) of MRX34 after IV dosing | 18 months
Number of patients with evidence of clinical activity of MRX34 | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: O'Neill VIncent, MD, Study Director — Mirna Therapeutics
Locations (10):
- United States (6):
  - Virginia G. Piper Cancer Center, Scottsdale, Arizona
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Texas Oncology Dallas, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Uthscsa/Ctrc, San Antonio, Texas
- South Korea (4):
  - Severance Hospital, Yonsie University Health System, Seoul, Seodaemun-Gu
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lucibello G, Mograbi B, Milano G, Hofman P, Brest P. PD-L1 regulation revisited: impact on immunotherapeutic strategies. Trends Mol Med. 2021 Sep;27(9):868-881. doi: 10.1016/j.molmed.2021.06.005. Epub 2021 Jun 26. PMID 34187739
- [Derived] Hong DS, Kang YK, Borad M, Sachdev J, Ejadi S, Lim HY, Brenner AJ, Park K, Lee JL, Kim TY, Shin S, Becerra CR, Falchook G, Stoudemire J, Martin D, Kelnar K, Peltier H, Bonato V, Bader AG, Smith S, Kim S, O'Neill V, Beg MS. Phase 1 study of MRX34, a liposomal miR-34a mimic, in patients with advanced solid tumours. Br J Cancer. 2020 May;122(11):1630-1637. doi: 10.1038/s41416-020-0802-1. Epub 2020 Apr 2. PMID 32238921